CLINICAL TRIAL: NCT05832216
Title: Efficacy of Daratumumab to Overcome Platelet Transfusion Refractoriness in Patients with Aplastic Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023015
Record Dates: First submitted 2023-04-03; First posted 2023-04-27 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Aplastic Anemia; Platelet Transfusion Refractoriness
Keywords: Platelet transfusion refractoriness; Daratumumab
MeSH Terms: conditions — Anemia, Aplastic | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daratumumab (Experimental)
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Daratumumab is a monoclonal globulin targeting the CD38 molecule of immune cells, which can eliminate antigen-presenting cells such as dendritic cells and macrophages, and indirectly reduce the production of autoantibodies. In addition, Daratumumab reduces autoantibody levels by targeting plasma cells, B lymphocytes and T lymphocytes.

SUMMARY:
This is a phase 1, prospective, single-arm, open-label study. The aim of this study is to evaluate the transfusion responses of platelet increment by using Daratumumab among aplastic anemia patients with platelet transfusion refractoriness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of aplastic anemia (AA)
* Dependent on platelet transfusions, characterized by either PLT<10×10^9/L, or PLT<20×10^9/L with bleeding events.
* Diagnosed with platelet transfusion refractoriness, characterized by Corrected count increment (CCI) <7500/ul at 60 min, or CCI <4500/ul at 24 hrs.
* Male or female age ≥ 12 years
* ECOG performance status ≤2
* Willing and able to comply with the requirements for this study and written informed consent.

Exclusion Criteria:

* The inherited bone marrow failure syndromes
* The presence of hemolytic PNH clone
* Combination of either radiotherapy or chemotherapy for solid tumors in recent 3 years, excluding the local tumor diagnosed 1 year ago and cured by surgical resection.
* Cytopenia caused by other diseases, including liver cirrhosis, active rheumatic connective tissue disease, and persistence of infectious diseases, etc.
* Uncontrolled infection
* HIV, HCV or HBV active infection
* The presence of any of the following bleeding events:

  * Gastrointestinal bleeding
  * Respiratory tract hemorrhage
  * Central nervous system bleeding
* Abnormal liver function: ALT or AST > 2 ULN, or TBil > 2 ULN after treatment.
* Abnormal kidney function: Creatinine clearance < 30 ml/min
* Heart failure (NYHA class III or IV)
* Poorly controlled diabetes, characterized by fasting blood glucose > 8.8mmol/L or post-meal blood glucose > 11.1mmol/L after therapy with insulin or oral hypoglycemic agents
* History of congestive heart failure, unstable angina pectoris, myocardial infarction, arterial or venous thrombosis
* Pregnant or breast-feeding patients
* Had a history of any psychiatric diseases, cerebrovascular disease or cognitive sequelae of head injury.
* Participation in another clinical trial within 4 weeks before the start of this trial
* Have an allergy to Daratumumab or any other part of this medicine.
* Previously treated with Daratumumab
* Previously treated with ATG/ALG within 4 months before the start of this trial
* Previously treated with the anti-CD20 monoclonal antibody within 2 months before the start of this trial
* Currently treated with TPO-RA except for a minimum of 4 weeks for washout before the start of this trial
* Patients considered to be ineligible for the study by the investigator for reasons other than above

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-10-12 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with platelet transfusion responsiveness | 12 weeks
  To evaluate the safety and efficacy of Daratumumab to increase the platelet increment, defined as Corrected Count Increment (CCI) ≥7500/μL at 60 min or CCI≥4500/μL at 24 hrs post transfusion, or platelet transfusion independence, i.e. PLT>10×10^9/L without any bleeding events.

SECONDARY OUTCOMES:
Time to the platelet increment | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Regenerative Medicine Center, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao Z, Pan H, Zhang L, Li W, Li R, Zhao J, Luo Y, Lian Y, Yu X, Kuang Z, Nie N, Li J, Huang J, Zhao X, Li Y, Fang L, Ge M, Zheng Y, Shi J. Targeting CD38 with daratumumab for platelet transfusion refractoriness in aplastic anemia. Blood. 2025 Jun 26;145(26):3189-3193. doi: 10.1182/blood.2025029006. PMID 40331918